CLINICAL TRIAL: NCT06728202
Title: A Horizontal Ridge Augmentation in Atrophic Maxillary Ridge: Evaluating Alveolar Ridge Splitting and Osseodensification
Brief Title: Osseodensification Versus Alveolar Ridge Splitting
Acronym: OD Vs ARS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Islam Wesam Saied Sayed, Administrative Dentist at Oral and Maxillofacial surgery department - Faculty of Dentistry at Fayoum University, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Horizontal Ridge Augmentation
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Maxillary Deficiency; Horizontal Alveolar Bone Defect
Keywords: Osseodensification; Alveolar Ridge Splitting; Dental implant
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized (1:1) clinical trial study formed of 2 competitive groups where 46 implants will be placed in 2 groups (23 for each group) to compare the Gained bone width in patients with atrophic maxillae (Horizontal defect) .
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alveolar ridge split group: (Active Comparator): * a crestal incision and two vertical releasing incisions will be formed, followed by a full-thickness mucoperiosteal flap.
  * the flap will be raised to expose the whole length facial cortical bone.
  * The palatal mucoperiosteum will also be slightly reflected for better exposure of the crest of the alveolar ridge and free placement of the surgical guides.
  * the patient specific guides will be placed and fixed by monocortical osteosynthesis screws at the pre-planned positions at the labial cortical plate of bone , precisely locate the mid-crestal and two vertical stop cuts to improve the accuracy of the procedure, preventing bad splits with the aim of reducing the final marginal bone loss associated with this technique.
  * bony cut will be performed using a piezoelectric device on the facial aspect of alveolar ridge 1.5 mm away from the adjacent teeth or implants, extending 7 mm apically from the crest of the ridge.implants will be inserted in the osteotomy sites using torque-wrench
  Interventions: Procedure: A Horizontal Ridge Augmentation in Atrophic Maxillary Ridge
- Implant placement in pristine bone with Osseodensification burs group: (Active Comparator): * A crestal incision and two vertical releasing incisions will be formed, followed by a full-thickness mucoperiosteal flap
  * Implant osteotomies are being performed with the assistance of saline irrigation. The osteotomies will be performed at 800-1500 rpm in a counterclockwise direction (Densifying Mode) with the use of sequential burs of similar diameter (OD drilling burs) used with copious irrigation in a Bouncing-Pumping motion (minor vertical pressure to advance the drill into the osteotomy, then pull out for pressure relief, then advance with vertical pressure again and so on in an in/out fashion). the instrumentation will be performed according to the recommended drilling protocols for Densah® Burs implant system; either by standard drilling, as recommended by implant company protocols.
  * The insertion of the implants will be initiated with the motor handpiece, without irrigation at 20-50 rpm, and installation will be completed with a manual surgical torque wrench
  Interventions: Procedure: A Horizontal Ridge Augmentation in Atrophic Maxillary Ridge

INTERVENTIONS:
Procedure: A Horizontal Ridge Augmentation in Atrophic Maxillary Ridge — Aiming to enhance bone volume (Quantity) in horizontal maxillary bone defects and density (Quality) , providing a viable solution for implant stability and long-term success.

SUMMARY:
Evaluation of clinical and radiological outcomes of the alveolar ridge splitting technique versus Osseodensification burs in atrophic maxillary alveolar ridges in horizontal dimension.

DETAILED DESCRIPTION:
The success of dental implant procedures hinges not only on the expertise of the clinician but also on the quality and quantity of bone at the implant site.

The significance of bone parameters in determining the feasibility and long-term outcomes of dental implants cannot be overstated. Over the years, various classifications have been proposed to assess bone quality and quantity, each aiming to provide a comprehensive framework for clinicians to evaluate and plan implant placement effectively.

One of the seminal classifications widely utilized in clinical practice is (the Cawood and Howell classification)1,2,3, which categorizes edentulous ridges into six types based on the quantity and quality of residual bone. In this classification system class IV in maxilla has gained special interest as it provides the adequate length for implant insertion but the width is insufficient. That made lots of researchers come with lots of different solutions to save time,cost and provide the best results for the patient.

Computed tomography (CT) provides an objective means to quantify bone density, expressed in Hounsfield units (HU), as described by T. Misch. The HU derived from CBCT scans correspond to grayscale values. Through linear regression analysis, grayscale values can be subjectively determined from CBCT images by aligning CT images with the same points on CBCT scans. The regression equation used for this analysis was HU = -61.098 + 1.178 × grayscale.4,5,6,7,8

Horizontal bone defects pose significant challenges in dental implantology, often requiring innovative surgical techniques to achieve successful implant placement.

Two emerging approaches, alveolar ridge splitting and osseodensification with specialized burs, have garnered attention for their potential in addressing such defects. These techniques aim to enhance bone volume (Quantity) and density (Quality) , providing a viable solution for implant stability and long term success.

1. Alveolar Ridge Splitting (ARST) :

   Alveolar ridge splitting, also known as horizontal or crestal osteotomy, is a surgical technique designed to increase the width of the alveolar ridge in cases of horizontal bone deficiency.

   The procedure involves carefully dividing the ridge and expanding it to create space for implant placement. Numerous studies have demonstrated the efficacy of ridge splitting in augmenting bone volume horizontally, allowing for the successful insertion of dental implants (Bassetti MA et al.2016)9.

   In a systematic review by Bassetti MA et al.2016 , alveolar ridge splitting was employed in patients with severe horizontal atrophy in the maxilla. The results indicated successful bone augmentation, with improved implant stability and survival rate.

   The technique exhibited minimal postoperative complications and demonstrated its potential as a reliable method for addressing maxillary horizontal bone defects.

   The ARST technique, by expanding buccal bone, prevents the dispersion of particulate bone substitutes and offers mechanical support against buccal mucosal tension. The expanded buccal bone also contains osteogenic stem cells and growth factors, potentially enhancing soft tissue healing and bone formation according to (Zhang L, Huang et al.2020)10 The systematic review conducted by (Elnayef B, Monje A et al.2015)11 and (Lin Y,Li G et al.2023)12 concluded that ARS technique: Predictable with high implant survival rate, adequate bone gain, and minimal complications and The weighted mean of horizontal bone width gain for full thickness flap ARS: 3.19 ± 1.19 mm (range: 2.00 to 4.03 mm)
2. Osseodensification Burs (OD) :

Osseodensification drilling protocol shows promise in cases of poor-quality autologous bone or challenging anatomical areas for implant stability. However, literature is limited, mainly comprising animal studies and short-term clinical cases. The technique's innovative nature necessitates specialized training for effective utilization according to (Inchingolo, A.D. et al.2021)13 Systematic Review. A study conducted by (Bergamo ETP et al., 2021)14 investigated the use of osseodensification burs in a series of cases involving maxillary horizontal bone atrophy. The results demonstrated improved primary implant stability and accelerated bone healing compared to traditional drilling techniques. Osseodensification not only addressed the bone defect but also facilitated faster osseointegration, contributing to successful implant outcomes.

A study conducted by (Koutouzis T et al., 2019)15 shows that the ridge dimensional percentage increase may reach up to 75% expansion in (3-4 mm) ridge width group.

Osseodensification not only addressed the bone atrophy, but also facilitated faster osseointegration, contributing to successful implant outcomes.x So Alveolar ridge splitting and osseodensification burs present promising solutions for maxillary horizontal bone defects, offering enhanced bone volume, density, and implant stability. Integrating these techniques into the treatment arsenal for implantology may provide clinicians with effective strategies to overcome the challenges posed by horizontal bone deficiencies in the maxilla.

ELIGIBILITY:
Inclusion Criteria:

I. Patients with atrophic maxillary alveolar ridges in horizontal dimension <18 years old. II. the bucco-palatal alveolar ridge dimension 2-4 mm III. a minimal vertical bone height of 10 mm

Exclusion Criteria:

I. Bad oral hygiene. II. Patients with non healthy habits as (Smokers, Alcoholics, or drug abusers). III. Patients with any active periapical pathosis. IV. Patients treated with chemo or radiotherapy during the past 5 years. V. Acute and progressive periodontal disease. VI. Medically compromised patient not indicated for surgical procedures. VII. Patient with history of bleeding disorders. VIII. Patient with osteo-porotic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Gained bone width : | preoperative , immediate postoperative and 6 months postoperative.
  will be measured immediately after surgery by CBCT using the following reference points:
  1. Ridge width (RW): the distance between the buccal and palatal border of the bone at the crest.
  2. Buccal bone thickness (BBT): the distance from the implant surface to the outer margin of bone. All variables will be measured twice with an interval of 1 week between measurements.

SECONDARY OUTCOMES:
Bone density : | Immediate post operative and 6 months postoperative
  CBCT to measure difference in bone density of newly formed bone at implant-crestal margin using the gray scale.
primary stability: | immediately and 6 months post-operative
  we measure using insertion Smartpeg specific for the implant system and restorative platform diameter will be used for each implant and perform a resonance frequency analysis using an OsstellMentor device18 (Ostell/Integration Diagnostics,Gothenburg, Sweden) to record ISQ19 values in all implant surfaces.

IPD SHARING:
Plan to Share IPD: Undecided